CLINICAL TRIAL: NCT03749200
Title: Clinical and Metabolic Efficacy of the Motivational Approach, Coordinated Between Primary Care and the Clinical Health Services for Childhood Obesity Treatment: Randomized Clinical Trial
Brief Title: Motivational Approach to Treat Childhood Obesity
Acronym: OBEMAT20
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: Institut Català de la Salut (Other); Hospital Universitari Joan XXIII de Tarragona. (Other); Hospital Universitari Sant Joan de Reus (Other); Instituto de Salud Carlos III (Other Government); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Ricardo Closa, Dr. PhD, Institut Investigacio Sanitaria Pere Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI15/00970
Record Dates: First submitted 2018-10-08; First posted 2018-11-21 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Childhood Obesity; Metabolic Syndrome; Body Composition
Keywords: Childhood Obesity; Motivational therapy
MeSH Terms: conditions — Pediatric Obesity; Metabolic Syndrome | interventions — Primary Health Care

STUDY DESIGN:
Intervention Model Description: Randomized clustered clinical trial, with treatment on obese children in 2 arms: a control group (CG) that will follow the usual recommendations of pediatricians and nurses in the primary care centres and an intervention group (IG) that will receive a structured motivation-based interview combined with group therapy and eHealth. the treatment of the two arms will last 12 (+3) months
Masking Description: Given the nature of the intervention participants or researchers could not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obemat2.0 Intervention Group (Experimental): Intervention: Obemat2.0 therapy (11 Motivational Interview Visits, 3 Workshops) Duration: 12 months (+3 months). Setting: Primary care centers Providers: pediatritians and nurses trained to perform motivational interview Visits description: The interviews follow a structure: 1. Checking the accomplishment of objectives to congratulate and motivate the patient. 2. A specific topic per visit is explained to the participant and family. 3. A task related to the topic (i.e. to plan a weekly menu for the family) is given to be brought back at the next visit. 4th. Objectives about diet, weight and physical activity are defined to be accomplished until the next visit. The follow-up of the structure is ensured by means of a printed material that the therapists provide each visit to participants.
  Interventions: Other: Obemat2.0 therapy
- Control Group (Active Comparator): Control Intervention: regular practise in primary care (11 individual monthly visits) Duration: 12 months (+3 months). Setting: Primary care centers. Providers: standard pediatritians and nurses Children and their families receive the usual recommendations conducted in primary care centers based on the Clinical Practice Guidelines on the Prevention and Treatment of Child and Adolescent Obesity. At visits, the family receive explanations about carrying out a balanced diet, divided into 5 meals, to provide a moderate energy reduction from the previous intake. An increase in physical activity, both in terms of leisure activity, as sports regular practise is recommended. Monthly visits are organized in which weight and height are measured and compliance with advice is reviewed.
  Interventions: Other: Regular practise in primary care

INTERVENTIONS:
Other: Obemat2.0 therapy
  Arms: Obemat2.0 Intervention Group
Other: Regular practise in primary care
  Arms: Control Group

SUMMARY:
The treatment of childhood obesity is challenging. Although dietary and physical activity recommendations are widely known, the willingness to change lifestyles within the family is not easy to be achieved. Motivational interviewing has been shown as a possibly effective method to increase adherence to dietary recommendations in the obese adult.

There is scarce evidence showing whether implementing a motivational interview in obese children could be effective.

The aim of this clinical trial is assessing the effect of a motivational interview, coordinated between the clinical and primary care services on 8 to 14 years old obese children.

DETAILED DESCRIPTION:
In a recent study, the investigators have demonstrated that the motivational therapy approach to treat childhood obesity is highly effective at clinical and metabolic levels. This efficacy has been proved in a clinical outpatient setting. However, a standardized collaborative approach between the clinic and the primary care services would allow a faster and easier approach to childhood obesity treatment. Furthermore, this motivational and educational intervention would benefit from the current technologic facilities, the long term effect of the education at group level, in terms of food shopping plan, healthy, fast and easy cooking methods.

The aim of this clinical trial is to test the efficacy of a multicomponent motivational intervention for the treatment of childhood obesity, coordinated between primary care and hospital specialized services, integrating motivational individual interviews, educational groups and eHealth tools (wearable), compared to the usual intervention performed in paediatrics.

The design will be a clustered randomized control trial, with an intervention group that will receive a multicomponent motivational and educational plan which will be compared to a control group receiving the usual recommendations performed in primary care centres (n=167 per group). The treatment of both study groups will last 12 months and will be performed at the primary care centres. In parallel, the study team will validate the methodology used to assess body composition in obese children as well as the changes produced by the intervention.

Children assigned to the control group receive advices as recommended by the Clinical Practice Guidelines (17). At visits, the family receive explanations about carrying out a balanced diet, divided into 5 meals, in order to provide a moderate energy intake reduction. An increase in physical activity, both in terms of leisure activity, as sports regular practise are recommended. Monthly visits are organized in which weight and height are measured, and compliance with recommendations are actually taking place.

Children assigned to the intervention group receive similar recommendations to those in the control group but under a motivational interview schema. This means that each visit, objectives from the last visit are fulfiled, the therapists try to make the family recongnizing the changes to be done by themselves, rather than imposing by demonstrating ambivalences, and objectives for the next visit are agreed. Furthermore, three workshops as group therapy are organized with the following topics: 1. Increasing physical actty sing an eHEalth monitor, 2. Food choices and dietary balance, and 3. Cooking methods.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 8 and <14 years at enrolment (so that, children would end the treatment at maximum age of 15 years
* BMI > 97th percentile of Hernandez references from 1988 (Hernández et al., 1988) as indicated by the Guidelines for Clinical Practice of the Spanish Health System (Grupo de trabajo de la Guía de Práctica Clínica sobre la Prevención y el Tratamiento de la Obesidad Infantojuvenil. Ministerio de Ciencia e Innovación [Spanish Ministry of Sciencee and Innovation], 2009) for the diagnose of the childhood obesity.

Exclusion Criteria:

* Children with eating disorders
* Families not available to attend to scheduled visits
* Simultaneous participation in another clinical trial
* Presence of endocrine disorders (GH disorder, hypothyroidism, Cushing's disease, early puberty or other)
* Lack of command of local languages

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 319 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Body Mass Index z-score | 12 (+3) months
  Changes in BMI z-score between the baseline visit and the final assessment

SECONDARY OUTCOMES:
Abdominal obesity (waist circumference) | 12 (+3) months
  Changes in waist circumference (cm) between the baseline visit and the final assessment
Abdominal obesity (waist to height) | 12 (+3) months
  Changes in waist-to-height circumference (ratio) between the baseline visit and the final assessment
Body composition: fat mass (kg) | 12 (+3) months
  Changes in fat mass (kg) between the baseline visit and the final assessment
Body composition: lean mass (kg) | 12 (+3) months
  Changes in lean mass (kg) between the baseline visit and the final assessment
Body composition: fat mass index (kg/m2) | 12 (+3) months
  Changes in fat mass index between the baseline visit and the final assessment
Body composition: lean mass index (kg/m2) | 12 (+3) months
  Changes in lean mass index between the baseline visit and the final assessment
HOMA-IR | 12 (+3) months
  Changes in insulin resistance between the baseline visit and the final assessment
Blood Pressure | 12 (+3) months
  Changes in systolic and diastoli blood pressure (s-score) between the baseline visit and the final assessment
Tryglycerides | 12 (+3) months
  Changes in tryglycerides (mg/dl) between the baseline visit and the final assessment

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Faculty of Medicine, C/ Sant Llorenç 21, Reus, Tarragona
  - Iispv- Hospital Sant Joan de Reus, Reus, Tarragona
  - IDIAP Jordi Gol, Reus, Tarragona
  - Hospital de Tarragona Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luque V, Feliu A, Escribano J, Ferre N, Flores G, Monne R, Gutierrez-Marin D, Guillen N, Munoz-Hernando J, Zaragoza-Jordana M, Gispert-Llaurado M, Rubio-Torrents C, Nunez-Roig M, Alcazar M, Ferre R, Basora JM, Hsu P, Alegret-Basora C, Arasa F, Venables M, Singh P, Closa-Monasterolo R. The Obemat2.0 Study: A Clinical Trial of a Motivational Intervention for Childhood Obesity Treatment. Nutrients. 2019 Feb 16;11(2):419. doi: 10.3390/nu11020419. PMID 30781525
- [Result] Luque V, Feliu A, Closa-Monasterolo R, Munoz-Hernando J, Ferre N, Gutierrez-Marin D, Guillen N, Basora J, Hsu P, Alegret-Basora C, Serrano MA, Mallafre M, Alejos AM, Balcells EN, Boada A, Paixa S, Mimbrero G, Gil-Mancha S, Tudela-Valls C, Alcazar M, Escribano J; Obemat2.0 Study Group. Impact of the motivational interviewing for childhood obesity treatment: The Obemat2.0 randomized clinical trial. Pediatr Obes. 2024 Jul;19(7):e13125. doi: 10.1111/ijpo.13125. Epub 2024 May 11. PMID 38733242
- See also: Results: access to full text — https://pubmed.ncbi.nlm.nih.gov/38733242/